CLINICAL TRIAL: NCT05252494
Title: The Effect Of Getting Children Between 3-6 To Watch Small Aquarium Fish On Physiological Parameters, Pain and Stress During Blood Collection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Tugba KARAKUS TURKER, Lecturer, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UskudarUskudar
Record Dates: First submitted 2022-01-11; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Bloodletting
Keywords: Pain management; animal assisted therapy; Aquarium Fish; Blood Collection; Physiological Parameters; Stress
MeSH Terms: conditions — Agnosia | interventions — Animal Assisted Therapy

STUDY DESIGN:
Intervention Model Description: The research consists of 2 groups as experimental and control group. In the experimental group, the children who watched the fish during the bloodletting process comprised the animal-assisted treatment group, and the control group consisted of the children who underwent routine bloodletting.
Who Masked: Participant
Masking Description: In this study, the Urn method, which is a randomization method equivalent to the full randomization method, will be used to determine the groups. In this randomization method, there are two parameters such as α and β. These parameters represent balls of two different colors, red and white. As a result of the lottery drawn in the research, the white ball will represent the "Animal assisted treatment group, and the red colored ball will represent the "Control Group". When there is a child who meets all the sampling criteria, the balls previously prepared by the researcher will be placed in a black bag and selection will be made by the nurse practitioner with their eyes closed. According to the color of the selected ball, it will be assigned to the child group, so that the children will be randomly distributed to the two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- animal assisted therapy group (Experimental): Animal assisted therapy group will watch aquarium fish while bloodletting prosedure.
  Interventions: Other: animal assisted therapy
- Control Group (No Intervention): Control group will not watch aquarium fish while bloodletting prosedure.

INTERVENTIONS:
Other: animal assisted therapy — In the intervention group, the child will be given to the mother's lap just before the invasive procedure. During the process, the aquarium with the fish will be placed on a shelf at a distance of about 50-60 cm, at an angle that the child can see. The camera on which the blood collection will be recorded will be placed on a tripod and placed on another shelf in such a way that the child can be seen completely. A video recording will be started 1 minute before the procedure, a pulse oximeter device will be attached to the child immediately after the child is seated on his mother's lap, physiological parameters, pain scores and stress will be determined. During the procedure, children's physiological measurements pain score and stress will be re-evaluated after the needle is inserted into the site. After the procedure, children's physiological measurements pain score and stress will be re-evaluated 1 minute after the needle is removed from the injection site
  Arms: animal assisted therapy group

SUMMARY:
Disease patterns are different from adults due to the fact that the abstract thinking and cause-effect abilities of children in the 3-6 age group are not developed. Children in this age group; Their ability to cope with stress is limited due to the need for special care, life experiences, mental development and inadequate ability to express themselves verbally (Conk et al, 2013). Illness is a source of pain and stress for them due to external factors and is a punishment for their bad behavior (Conk et al, 2013; Teksöz & Ocakçı, 2014).Hospital, on the other hand, means foreign environment/persons, loss of independence, loss of privacy, painful procedures, disruption of daily routines, surgery, pain, disability, death, separation from family and friends for children (Conk et al, 2013). Blood collection and vascular access are the interventions that cause the most pain, stress and anxiety in hospitalized children (Duff, 2003; Caprilli et al, 2007) . Non-invasive non-pharmacological methods increase the release of endorphins, the body's natural morphine, and relieve pain, thereby reducing the stress and anxiety of the child and family (Bergomi et al, 2018). Clinical experience argues that human-animal bonding, which is one of the distraction practices in pain management, is effective in reducing pain and stress (Muslu, 2011; Min & Zaw 2016; Alvarez et al, 2020) .

In the light of all this information; The aim of this study was to determine the effect of watching small aquarium fish, which is used as a distraction method during the blood collection process, on the pain and stress, heart rate and oxygen saturation during the procedure in children aged 3-6 years who applied to the blood collection unit.

Hypotheses of the Research:

Hypothesis 0 (H0): Feelings felt by children watching and not watching fish during blood collection there was no difference between stress, pain score, heart rate, oxygen saturation, crying and procedure time.

Hypothesis 1 (H1): The oxygen saturation of the children who watched the fish during the blood collection process is high.

Hypothesis 2 (H2): Children watching the fish during the blood draw have a higher heart rate is low.

Hypothesis 3 (H3): Children who watched the fish during the blood draw had a higher pain score is low.

Hypothesis 4 (H4): The stress score of the children who watched the fish during the blood collection process was higher is low.

Hypothesis 5 (H5): The crying time of the children watching the fish during the blood collection process is longer is short.

Hypothesis 6 (H6): The processing time is longer for children watching the fish during the blood collection process is short.

DETAILED DESCRIPTION:
The universe of the research will be all children brought to a training and research hospital for blood transfusion between March 2022 and March 2023. The sample of the study will be the children of parents who comply with the sample selection criteria and volunteer to participate in the research.

In order to determine the number of samples, power analysis was performed using the G*Power (v3.1.7) program. The power of the study is expressed as 1-β (β = probability of type II error), and in general studies should have 80% power. Based on the pain measurement differences before and after the procedure in Carie Braun's study to evaluate the pain during blood collection (difference of the means for the control group: 0.31; the difference of the mean for the experimental group was 1.61), the effect size was calculated to obtain 80% power at the α=0.05 level. (d) 0.748 was found. According to this, it was calculated that there should be at least 30 people in each group and 60 people in total. Considering that there may be losses during the study process, it was decided to take at least 35 people in each group.

Data Collection Tools and Materials: The following tools and forms will be used in the collection of research data: Informed Voluntary Consent Form (Appendix 1): Before starting the research, all children's parents should be informed about the purpose, plan, duration of the research, how the obtained data will be used "Voluntary Information and Consent Form" " and verbal and written permissions will be obtained. Parents who agree to participate in the study will be told that they can withdraw from the study at any time, they will be assured that the individual information obtained will not be disclosed to anyone other than the researcher, and that no fees will be charged to the parents or that no research expense will be charged to the social security institution to which the patient is affiliated.

Information Form (Appendix 2): It was prepared by scanning the literature on the subject. The information form is the form in which the child's name, surname, group, introductory information about the parents and the child are recorded. The information form will be filled by the researcher himself by face-to-face interview method. Follow-up Form (Appendix 3): It was prepared by scanning the literature on the subject. The follow-up form is the form in which the child's pain and stress score, physiological parameters, crying and duration of the procedure are recorded. The follow-up form will be filled in by the researcher himself in line with the findings obtained from the patient during data collection.

Pain Assessment Tool (FLACC) (Appendix 4):

It was developed by Merkel (1997), and Turkish validity and reliability was done by Şenaylı et al (2006). Each of the baby's facial expression, leg movements, activity, crying and comfortability parameters consists of three sub-items and can be applied to children aged 1 month to 9 years. The items take the value 0, 1, 2, respectively, and the total score is between 0 and 10. A "0" score indicates no pain, 1-3 points mild, 4-6 points moderate and 7-10 points severe pain. In order to use the FLACC pain assessment scale, permission was obtained from Şenaylı et al. via e-mail.

Wong and Baker Faces Pain Scale [Wong-Baker Faces Pain Rating Scale (WBFPRS) (Appendix 5): This scale was developed by Donna Wong and Connie Morain Baker in 1988. This scale is used to diagnose pain in children aged 3-18 years. Studies comparing this tool with others have reported that children like the facial expressions rating scale and that it provides the most accurate pain measurement. In this scale, pain scores are given according to the numerical values given to the faces. The lowest score is "1" and the highest score is "5". As the score obtained from the scale increases, the pain tolerance decreases, and as the score decreases, the tolerance increases.

Children's Emotional Manifestation Scale-CEMS (Appendix 6): Children's Emotional Expression Evaluation Scale; The scale, which was developed by Ho Cheung William Li (Children's Emotional Manifestation Scale-CEMS) in 2003 and validated in Turkish by Yanık and Ark (2019), consists of a total of 5 different categories and 25 items. This scale evaluates the anxiety experienced by children during medical procedures. In the facial expression category of the first 5 items, the facial expressions of the child observed by the researcher are scored. Secondly, the child's tear state is evaluated over 5 sub-items in the vocalization category. Third, in the 5 sub-items of the movement title, the child's body language is scored. Fourth, the child's verbal or non-verbal communication is evaluated in 5 sub-items in the interaction category. Fifth, scoring is done by observing the active or passive participation of the child in the 5 sub-items of the cooperation category. 1-5 points in each category

ELIGIBILITY:
Inclusion Criteria:

* Parents' willingness to participate in the research is in line with the voluntary consent form have obtained written consent from their parents,
* The child is between 3-6 years old,
* The child musn't not have fish,
* No blood sampling has been performed in the last year,
* If the child is considered healthy as a result of the examination performed by the doctor,

Exclusion Criteria:

* if The child has fish
* To have taken analgesic medication 4 hours before the procedure
* if The child is afraid of fish,
* The child has a known allergy history,
* Deterioration of skin integrity in the blood collection area,
* ifThe child has a visual/hearing disability.
* if The child has developmental delay, mental problems
* if there is Failure of blood collection in the first attempt.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Differences in physiological parameters | 1 year
  Differences in oxygen saturation
Differences in physiological parameters | 1 year
  Differences in heart rate
Differences in pain score | 1 year
  Pain Assessment Tool (FLACC):
  The items take the value 0, 1, 2, respectively, and the total score is between 0 and 10. A "0" score indicates no pain, 1-3 points mild, 4-6 points moderate and 7-10 points severe pain.
Differences in pain score | 1 year
  Wong and Baker Faces Pain Scale [Wong-Baker Faces Pain Rating Scale (WBFPRS): The lowest score is "1" and the highest score is "5". As the score obtained from the scale increases, the pain tolerance decreases, and as the score decreases, the tolerance increases.
Differences in stress | 1 year
  Children's Emotional Manifestation Scale-CEMS: Scale consists of a total of 5 different categories and 25 items. As the score obtained from the scale increases, the pain tolerance decreases, and as the score decreases, the tolerance increases.
Differences in crying time | 1 year
  Crying time will be measured by chronometer (second/minute)
Differences in procedure time | 1 year
  Prosedure time will be measured by chronometer (second/minute)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teksöz, E. Ocakçı, A. F. Çocuk Hemşireliği'nde Sanat Uygulamaları. Dokuz Eylül Üniversitesi Hemşirelik Fakültesi Dergisi.2014; 7(2): 119- 123.
- [Background] Duff AJ. Incorporating psychological approaches into routine paediatric venepuncture. Arch Dis Child. 2003 Oct;88(10):931-7. doi: 10.1136/adc.88.10.931. PMID 14500318
- [Background] Bergomi P, Scudeller L, Pintaldi S, Dal Molin A. Efficacy of Non-pharmacological Methods of Pain Management in Children Undergoing Venipuncture in a Pediatric Outpatient Clinic: A Randomized Controlled Trial of Audiovisual Distraction and External Cold and Vibration. J Pediatr Nurs. 2018 Sep-Oct;42:e66-e72. doi: 10.1016/j.pedn.2018.04.011. Epub 2018 May 1. PMID 29728296
- [Background] Caprilli S, Anastasi F, Grotto RP, Scollo Abeti M, Messeri A. Interactive music as a treatment for pain and stress in children during venipuncture: a randomized prospective study. J Dev Behav Pediatr. 2007 Oct;28(5):399-403. doi: 10.1097/DBP.0b013e31811ff8a7. PMID 18049324
- [Background] Muslu, G. K. Conk, K. Hayvan Destekli Uygulamalar Ve Çocuklarda Kullanımı. Deuhyo Ed 2011, 4 (2), 83-88.
- [Background] Min, M. Zaw, C.C. A Review On Animal-Assisted Therapy And Activities For Healthcare And Teaching Of Children. Journal Of Education And Social Sciences.2016;(3), 40-46.
- [Background] Avila-Alvarez A, Pardo-Vazquez J, De-Rosende-Celeiro I, Jacome-Feijoo R, Torres-Tobio G. Assessing the Outcomes of an Animal-Assisted Intervention in a Paediatric Day Hospital: Perceptions of Children and Parents. Animals (Basel). 2020 Oct 1;10(10):1788. doi: 10.3390/ani10101788. PMID 33019696
- [Background] Conk Z, Başbakkal Z, Bal Yılmaz H, Bolışık B. Pediatri Hemşireliği. Akademisyen Tıp Kitabevi, Ankara, 2013.
- [Background] Braun C, Stangler T, Narveson J, Pettingell S. Animal-assisted therapy as a pain relief intervention for children. Complement Ther Clin Pract. 2009 May;15(2):105-9. doi: 10.1016/j.ctcp.2009.02.008. Epub 2009 Mar 3. PMID 19341990
- [Background] Yanık, M. Kuzlu Ayyıldız, T. Kulakçı Altıntaş, H. Çocukların Duygusal Dışa Vurumunu Değerlendirme Ölçeği: Geçerlik Ve Güvenirlik Çalışması. Anadolu Hemşirelik Ve Sağlık Bilimleri Dergisi, 2019; 22(3): 179-188
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Şenaylı, Y. Özkan, F. Şenaylı, A. Bıçakçı, Ü. Çocuklarda Postoperatif Ağrının FLACC (YBAAT) Ağrı Skalasıyla Değerlendirilmesi. Turkiye Klinikleri J Anest Reanim. 2006;4(1):1-4
- [Background] Wong DL, Baker CM. Pain in children: comparison of assessment scales. Pediatr Nurs. 1988 Jan-Feb;14(1):9-17. No abstract available. PMID 3344163